CLINICAL TRIAL: NCT05697237
Title: Exploratory Clinical Study of Carlizumab Plus Sovantinib in Second-line Treatment of Advanced or Metastatic Cholangiocarcinoma
Brief Title: Carlizumab Plus Sovantinib in Second-line Treatment of Advanced or Metastatic Cholangiocarcinoma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XJTU1AF2021LSK-368
Record Dates: First submitted 2022-12-21; First posted 2023-01-25 (Actual); Last update posted 2023-01-25 (Actual); Status verified 2022-12

CONDITIONS: Cholangiocarcinoma
MeSH Terms: conditions — Cholangiocarcinoma | interventions — camrelizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Advanced or metastatic cholangiocarcinoma (Experimental): In this study, carrilizumab combined with sovantinib in the second-line treatment of patients with advanced or metastatic cholangiocarcinoma with single arm, open, Exploratory clinical trials.The specific treatment regimen was carrilizumab 200mg Q3W d1; Sofantinib: 300mg,Take orally, once a day, continuously. Treatment continues or until disease progression occurs or the patient becomes intolerant to treatment regimens.The efficacy was evaluated every 2 cycles.
  Interventions: Drug: Carrelizumab; Drug: Solfantinib

INTERVENTIONS:
Drug: Carrelizumab — Carrelizumab 200mg/3 weeks
Drug: Solfantinib — Solfantinib 300mg/d

SUMMARY:
The incidence of cholangiocarcinoma is high, the radical resection rate is low, the postoperative recurrence is easy, the prognosis is poor.Gemcitabine combined with cisplatin (GC) is the standard first-line treatment for patients with advanced biliary carcinoma, and up to now there is no standard second-line treatment Commend.Carrilizumab was highly effective in previous studies,Its combined GEMOX protocol has been published in the "Guidelines for the Diagnosis and Treatment of Gallbladder Cancer (2019 Edition)" and the "China Clinical Oncology" The Society's (CSCO) Guidelines for the Diagnosis and Treatment of Biliary alignancies 2020 is recommended for the first-line treatment of advanced biliary cancers.Solfantinib is targeted at VEGFR1, 2, 3, FGFR1And CSF1R highly selective small molecule targeted therapy drugs. Data from a preliminary phase 2 clinical trial observed sofantinib therapy Survival benefits of cholangiocarcinoma patients in China.

DETAILED DESCRIPTION:
In this study, carrilizumab combined with suvantinib in the second-line treatment of patients with advanced or metastatic cholangiocarcinoma with single arm, open, Exploratory clinical trials. The study plan enlists 60 patients with unresectable or recurrent disease confirmed by histopathology or cytology Or metastatic cholangiocarcinoma (including intrahepatic cholangiocarcinoma, extrahepatic cholangiocarcinoma, distal cholangiocarcinoma). Past acceptance of standard containing Systematic internal medicine anti-tumor therapy with gemcitabine regimen met the inclusion criteria of this study, and carrilizumab combined with cord was given Vantinib oral therapy. The specific treatment regimen was carrilizumab 200mg Q3W d1; Solventinib: 300mg, Orally, once a day, continuously. Treatment continues or until disease progression occurs or the patient becomes intolerant to the treatment regimen The efficacy was evaluated every 2 cycles. The main evaluation of carrilizumab combined with suvantinib in second-line treatment was advanced or Progression-free survival (PFS) in patients with metastatic cholangiocarcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. Advanced inability to root was pathologically confirmed Patients with curatively resected or metastatic bile duct epithelial cell carcinoma;
2. had previously received systemic antitumor therapy with a chemotherapy regimen (including gemcitabine)
3. Age ≥18 and under 75
4. Predicted survival ≥3 months
5. ECOG score 0-1
6. Child-Pugh score < 8
7. There was at least one measurable tumor lesion with a long diameter ≥10 mm and a short diameter ≥15 mm on spiral CT，For general CT or physical examination, the maximum diameter must be ≥20mm
8. The results of liver and kidney function and blood routine examination within 1 week before enrollment were consistent with the following conditions：ANC≥1.5×10^9/L,PLT≥80×10^9/L,HGB≥80g/L,Cr≤1.5×ULN,TBIL≤2.5×ULN,ALP≤2.5×ULN,AST≤2.5×ULN,ALT≤2.5×ULN
9. Patients participate voluntarily and sign informed consent forms

Exclusion Criteria:

1. Known allergies to carrilizumab or solfantinib machine components
2. Patients with obstructive jaundice who could not reach the upper limit of TBIL≤2.5 times of normal value after surgical intervention
3. Patients with biliary obstruction that may occur or worsen within 4 to 6 weeks
4. Patients with obvious coagulation mechanism disorder, active bleeding and bleeding tendency
5. History of other malignancies within 5 years (fully treated basal cell carcinoma of the skin, cervical cancer in situ)
6. Interstitial pneumonia or pulmonary fibrosis
7. Uncontrollable pleural effusion or ascites
8. Severe uncontrolled medical disease, acute infection, recent history of myocardial infarction (within 3 months)
9. Pregnant or lactating mothers who refused to take appropriate contraceptive measures during the course of the study;
10. The researchers determined that the patients were not suitable for this study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-01 (Estimated); Primary Completion 2024-06 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
PFS | 6months
  Progression Free Survival

SECONDARY OUTCOMES:
ORR | 6months
  Objective Response Rate
OS | 12months
  Overall Survival
DCR | 6months
  Disease control rate Disease control rate Disease control rate

CONTACTS AND LOCATIONS:
Overall Officials: enxiao li, PHD, Principal Investigator — First hospital of Xi'an Jiaotong University